CLINICAL TRIAL: NCT06086977
Title: Pulse Analysis for Cholecystitis Patients Before and After Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Taichung Tzu Chi Hospital (Other)
Responsible Party: Principal Investigator, I-Hsuan Chien, Doctor of Chinese medicine department, Principal Investigator, Resident physician, Taichung Tzu Chi Hospital
Other Study IDs: REC110-12
Record Dates: First submitted 2022-09-22; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Cholecystitis; Cholecystectomy
Keywords: radial pressure pulse (RPP)
MeSH Terms: conditions — Cholecystitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to record the radial pressure pulse(RPP) of the patients with cholecystitis compared preoperative and postoperative pulse changes in an attempt to determine the relationship between cholecystitis and pulse.

DETAILED DESCRIPTION:
A total of 20 patients were recruited according to the inclusion and exclusion criteria. The patients, aged 32-76 years, were given a diagnosis of cholecystitis by a general surgeon from Taiwan's Taichung Tzu Chi Hospital. All eligible patients included in the study agreed to participated and signed the informed consent form and the study procedures were approved by the ethical committee of Taichung Tzu Chi general hospital (REC110-12). By measuring and recording the RPP preoperatively and postoperatively, the mean values of the spectral energy (SE0-10 Hz, SE10-50 Hz, and SE13-50 Hz) were obtained for comparison with the preoperative white blood cell (WBC) count.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with acute or chronic cholecystitis
2. Patient hospitalized for cholecystectomy
3. Patients who were voluntarily involved in this study

Exclusion Criteria:

1. Patients who could not cooperate with pulse diagnosis
2. Patients with underlying systemic diseases such as cancer, chronic obstructive pulmonary disease, cardiac failure, chronic renal failure, cirrhosis, etc.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cholecystitis and recieve cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-02-12 (Actual); Study Completion 2022-06-12 (Actual)

PRIMARY OUTCOMES:
The changes of spectral energy of radial artery pulse after cholecystectomy | Baseline (before cholecystectomy) and 24 -48 hours after cholecystectomy
  The spectral energy of radial artery pulse was measured before and after cholecystectomy to compare the difference

CONTACTS AND LOCATIONS:
Locations (1):
- TZU CHI Hospital, Taichung, Taiwan